CLINICAL TRIAL: NCT05628441
Title: Real-time Computer Aided Detection of Barrett's Neoplasia: a Pilot Study
Brief Title: Real-time Computer Aided Detection of Barrett's Neoplasia
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, prof. dr. J.J.G.H.M. Bergman, Professor of Gastroenterology, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2021.0269
Record Dates: First submitted 2022-10-28; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Barrett Esophagus; Barrett Adenocarcinoma
Keywords: Barrett's Esophagus; Computer Aided Detection
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CADe system: All patients included in the study will undergo the endoscopic procedure according to standard clinical care and the study protocol. The CADe system will run in the back, not interfering with care.
  Interventions: Other: Computer Aided Detection system for Barrett's neoplasia

INTERVENTIONS:
Other: Computer Aided Detection system for Barrett's neoplasia — CADe system running in the back, not directly interfering with patient care

SUMMARY:
In the real-time pilot study, the performance of a recently developed Computer Aided Detection (CADe) system will be investigated in 30 patients during real-time live endoscopic examination. Three expert endoscopists in the field of Barrett's esophagus and endoscopic resection techniques will perform the inclusions following a standardized data acquisition protocol. In total, 15 patients with a visible neoplastic lesion in their Barrett's esophagus and 15 patients without any visible abnormalities in their Barrett's esophagus will be included in this study. Outcomes: to investigate feasibility of the use of the CADe system in the endoscopy suite, to investigate the performance of the CADe system when used by endoscopists.

DETAILED DESCRIPTION:
Patients in this study will undergo a scheduled surveillance endoscopy (according to current guidelines; n = 15) or are referred to a tertiary referral center for endoscopic resection of a possible neoplastic area in their known Barrett's esophagus (n = 15).

Patients will be consciously sedated (standard care) before start of the procedure. During the endoscopic procedure, the endoscopist follows the standard protocol after extensive cleaning of the Barrett's segment: first, a standardized pullback video will be recorded, followed by a careful inspection of the Barrett segment every 2 centimeters. Per 2cm, a video of 10 seconds and 3 overview images are being recorded.

During the imaging protocol, the CADe system presents its prediction on a second screen, next to the main endoscopy monitor. After the imaging protocol, standard clinical care is being resumed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patients under surveillance for their diagnosed non-dysplastic Barrett's esophagus or patients refered for endoscopic treatment because of proven high-grade dysplasia or adenocarcinoma;
* A circumferential Barrett length of at least 2cm

Exclusion Criteria:

* Medical history of prior surgical or endoscopical treatment for neoplasia in their esophagus
* Reflux esophagitis > grade 2 (LA classification)
* Inability to undergo endoscopic treatment and/or biopsies

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Barrett's esophagus, either receiving a surveillance endoscopy according to protocol or referred for endoscopic treatment for proven neoplasia in their Barrett's esophagus
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Combined performance of endoscopist + CADe system in terms of per-patient sensitivity and specificity | 5 months
  To investigate the combined performance between endoscopist and CADe system on a per-patient level.

SECONDARY OUTCOMES:
Stand-alone performance of CADe system in terms of per-patient sensitivity and specificity | 5 months
  To investigate the performance of the CADe system on new data on a per-patient level.

CONTACTS AND LOCATIONS:
Overall Officials: J.J. Bergman, MD PHD, Principal Investigator — Amsterdam University Medical Centers, location AMC
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared

REFERENCES:
- [Derived] Fockens KN, Jukema JB, Jong MR, Boers T, van der Putten JA, Kusters CHJ, Pouw RE, Duits LC, van der Sommen F, de With PH, de Groof AJ, Bergman JJ; BONS-AI consortium. The use of a real-time computer-aided detection system for visible lesions in the Barrett's esophagus during live endoscopic procedures: a pilot study (with video). Gastrointest Endosc. 2024 Sep;100(3):527-531.e3. doi: 10.1016/j.gie.2024.04.011. Epub 2024 Apr 9. PMID 38604297